CLINICAL TRIAL: NCT03915847
Title: Evaluation of Cesarean Scar After Three Different Uterine Closure Technis: A Randomised Trial
Brief Title: Evaluation of Cesarean Scar After Three Different Uterine Closure Technis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ragıp Atakan Al, Proffesor in dept. of obstetrics and gynecology, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATA35
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Cesarean Section, Repeated; Cesarean, Uterine Scar Thickness; Cesarean, Residual Myometrial Thickness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single layer closure (Active Comparator)
  Interventions: Procedure: Single layer closure
- Double layer closure (Active Comparator)
  Interventions: Procedure: Double layer closure
- Doble layer closure with trimming (Active Comparator)
  Interventions: Procedure: Doble layer closure with trimming

INTERVENTIONS:
Procedure: Single layer closure — Uterine incision will be approximated with continuous unlocked suture, including a narrow band of the endometrial layer, without trimming incision edges.
  Arms: Single layer closure
Procedure: Double layer closure — The first layer suture penetrated the whole thickness of the uterine wall, including a narrow band of the endometrial layer. Second layer sture is acontinous sture performed in a lateral-to lateral position , imbricating first layer.
  Arms: Double layer closure
Procedure: Doble layer closure with trimming — Uterine incision will be trimmed and old scar tissue will be removed. The first layer suture penetrated the whole thickness of the uterine wall, including a narrow band of the endometrial layer. Second layer sture is acontinous sture performed in a lateral-to lateral position , imbricating first layer.
  Arms: Doble layer closure with trimming

SUMMARY:
The study compares three techniques of uterine closure on myometrium thickness at the site of uterine scar of women who underwent repeated cesarean section. Cesarean scar will be evaluated by transvaginal ultrasound six months after cesarean.

ELIGIBILITY:
Inclusion Criteria:

* Previous two or three cesarean
* Gestational weeks >=36 weeks

Exclusion Criteria:

* Risk of obstetric haemorrhage
* Suspicion or diagnosis placenta previa or accrete syndrome
* Chorioamnionitis
* Uterine myoma in the anterior uterine segment
* Hysterotomy other than lower segment uterine incision at previous cesarean

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Residual myometrial thickness | 6 months after cesarean
  Myometrial thickness at the uterine scar by transvaginal ultrasound

SECONDARY OUTCOMES:
Existence of cesarean scar defect | 6 months after cesarean
  The presence or absence of a cesarean scar defect that was defined as any unechogenic area visualised by transvaginal ultrasound at the site of the cesarean scar with a depth of at least 2 mm.
Width of defect | 6 months after cesarean
  In a sagittal plane, the width at base of defect
Depth of defect (niche) | 6 months after cesarean
  In a sagittal plane, the distance from the base lining of the endometrium to the apex
Operation time | 10 minute after cesarean completed
  Skin-to-skin operation time
Change in hemoglobin | 48 hours after cesarean
  Difference in haemoglobin measured preoperatively and postoperatively 48 hours
Blood product transfusion | One week after cesarean
  Unite number of transfused packed erythrocyte
Maternal infectious morbidity | Six weeks after cesarean
  Prevalence of postpartum endometritis, skin wound dehiscence and post operative fever.
Length of hospitalization | One month after cesarean
  Duration in days

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)